CLINICAL TRIAL: NCT00510874
Title: A Phase I/II, Observer-Blind, Randomized, Active-Controlled Trial to Evaluate the Safety and Immunogenicity of a Two-Dose Series of GSK Biologicals' Candidate Influenza Vaccine GSK 1557484A Antigens With or Without Adjuvant
Brief Title: Study to Evaluate the Safety and Immune Response of Two-Doses of Candidate Influenza Vaccine GSK 1557484A in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110028
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza; GSK 1557484A vaccine
MeSH Terms: conditions — Influenza, Human | interventions — pandemrix

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Pumarix Formulation 1 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 1 of Pumarix™ vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
  Interventions: Biological: Pumarix™
- Pumarix Formulation 2 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 2 of Pumarix™ vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
  Interventions: Biological: Pumarix™
- Pumarix Formulation 3 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 3 of Pumarix™ vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
  Interventions: Biological: Pumarix™
- Pandemrix Formulation A Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation A of Pandemrix™ vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
  Interventions: Biological: Pandemrix ™
- Pandemrix Formulation B Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation B of Pandemrix ™ vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
  Interventions: Biological: Pandemrix ™
- Pumarix Formulation 4 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 4 of Pumarix™ vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
  Interventions: Biological: Pumarix™
- Pumarix Formulation 5 Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 5 of Pumarix™ vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
  Interventions: Biological: Pumarix™

INTERVENTIONS:
Biological: Pumarix™ — Two doses administered intramuscularly (IM), the first in the deltoid region of the non-dominant arm and the second in the deltoid region of the dominant arm.
  Arms: Pumarix Formulation 1 Group; Pumarix Formulation 2 Group; Pumarix Formulation 3 Group; Pumarix Formulation 4 Group; Pumarix Formulation 5 Group
Biological: Pandemrix ™ — Two doses administered intramuscularly (IM), the first in the deltoid region of the non-dominant arm and the second in the deltoid region of the dominant arm.
  Arms: Pandemrix Formulation A Group; Pandemrix Formulation B Group

SUMMARY:
The purpose of this study is to evaluate the safety and immune response of two-doses of GSK Biologicals' candidate influenza vaccine GSK 1557484A with or without adjuvant in adults. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The study has five core arms and the stratification is based on site and age. In addition, there are 4 possible contingent groups of which 2 will be studied based on an analysis concerning immunogenicity performance at Day 42 in core groups above.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults 18 to 64 years of age at time of first vaccination, inclusive.
* Good general health as assessed by medical history and physical examination.
* Access to a consistent means of telephone contact
* Written informed consent obtained from the subject.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.

Exclusion Criteria:

* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Blood pressure abnormalities
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and may enroll, but other histologic types of skin cancer are exclusionary.
* Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylactic tamoxifen are excepted and may enroll.
* Presence of an oral temperature ≥ 37.8º C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of cytotoxic or immunosuppressive drug within 6 months of study enrollment.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin.
* Administration of any non-influenza vaccines within 30 days before study enrollment or during the study period.
* Use of any investigational or non-registered product (drug or vaccine) or planned participation in another investigational study within 30 days prior to study enrollment, or during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrollment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (ß-hCG) test result prior to dosing on Study Days 0 or 21.
* Lactating or nursing.
* Women of child bearing potential who lack a history of reliable contraceptive practices.
* Known receipt of analgesic or antipyretic medication on the day of treatment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 780 (Actual)
Dates: Start 2007-07-28; Primary Completion 2008-06-17 (Actual); Study Completion 2008-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (7):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Las Vegas, Nevada
- Canada (3):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Langley JM, Frenette L, Ferguson L, Riff D, Sheldon E, Risi G, Johnson C, Li P, Kenney R, Innis B, Fries L. Safety and cross-reactive immunogenicity of candidate AS03-adjuvanted prepandemic H5N1 influenza vaccines: a randomized controlled phase 1/2 trial in adults. J Infect Dis. 2010 Jun 1;201(11):1644-53. doi: 10.1086/652701. PMID 20423222
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 110028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110028 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Started | 78 | 152 | 151 | 151 | 148 | 50 | 50
Completed | 75 (Upto Day 182) | 148 (Upto Day 182) | 150 (Upto Day 182) | 148 (Upto Day 182) | 141 (Upto Day 182) | 50 (Upto Day 182) | 49 (Upto Day 182)
Not Completed | 3 | 4 | 1 | 3 | 7 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 1 | 3 | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group | Total
Number analyzed (Participants) | 78 | 152 | 151 | 151 | 148 | 50 | 50 | 780
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.5 (12.85) | 38.1 (12.10) | 39.0 (12.59) | 38.7 (11.25) | 38.7 (12.20) | 39.2 (12.21) | 39.9 (13.18) | 38.8 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 83 | 87 | 100 | 78 | 32 | 24 | 449
  Male | 33 | 69 | 64 | 51 | 70 | 18 | 26 | 331

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer on the specified day.
Time Frame: At Day 42
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data for the primary outcome variables were available i.e. all subjects had to have at least Day 0 and Day 42 HI titer results for the A/Indonesia/5/05 virus.
Measure: Count of Participants; unit: Participants
Groups:
- Pumarix Formulation 1 Group: Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 1 of Pumarix vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
- Pumarix Formulation 2 Group: Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 2 of Pumarix vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
- Pumarix Formulation 3 Group: Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 3 of Pumarix vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
- Pandemrix Formulation A Group: Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation A of Pandemrix vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
- Pandemrix Formulation B Group: Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation B of Pandemrix vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
- Pumarix Formulation 4 Group: Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 4 of Pumarix vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
- Pumarix Formulation 5 Group: Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of formulation 5 of Pumarix vaccine at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm (non-dominant arm for the first injection and dominant arm for the second one).
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 75 | 144 | 146 | 140 | 142 | 49 | 50
Participants | 13 | 140 | 131 | 135 | 131 | 47 | 42

2. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 75 | 144 | 146 | 140 | 142 | 49 | 50
Titers | 10.5 [8.2 to 13.5] | 464.7 [383.4 to 563.4] | 320.7 [246.9 to 416.6] | 480.3 [390.5 to 590.7] | 347.7 [272 to 444.5] | 331.6 [217.4 to 505.6] | 173.9 [105.6 to 286.3]

3. Primary Outcome: Number of Seroprotected Subjects Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 75 | 144 | 146 | 140 | 142 | 49 | 50
Participants | 13 | 140 | 131 | 135 | 131 | 47 | 42

4. Primary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any solicited local symptoms regardless of their intensity grade. Any redness and swelling were ≥ 20 millimeters (mm).
Time Frame: Within the 7-day follow-up period (Days 0-6) after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who received at least one dose of vaccine for whom any post-vaccination data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 78 | 152 | 151 | 151 | 148 | 50 | 50
Participants
  Any Pain | 18 | 133 | 130 | 139 | 124 | 48 | 42
  Any Redness | 0 | 7 | 2 | 9 | 6 | 1 | 0
  Any Swelling | 0 | 12 | 10 | 21 | 9 | 4 | 0

5. Primary Outcome: Number of Subjects With Solicited General Symptoms.
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location (joint pain), muscle aches, shivering, sweating and fever. Fever was defined as oral temperature (≥) 38 degrees Celsius (°C). Any = occurrence of any solicited general symptoms regardless of intensity grade or relationship to vaccination.
Time Frame: Within the 7-day follow-up period (Days 0-6) after any vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 78 | 152 | 151 | 151 | 148 | 50 | 50
Participants
  Any Fatigue | 16 | 64 | 50 | 67 | 69 | 15 | 15
  Any Headache | 25 | 71 | 61 | 66 | 61 | 11 | 19
  Any Joint Pain | 12 | 49 | 36 | 53 | 39 | 11 | 11
  Any Muscle Aches | 15 | 74 | 64 | 86 | 63 | 19 | 21
  Any Shivering | 4 | 18 | 21 | 27 | 17 | 8 | 6
  Any Sweating | 6 | 23 | 12 | 24 | 21 | 5 | 1
  Any Fever | 0 | 4 | 3 | 12 | 11 | 1 | 0

6. Primary Outcome: Number of Subjects With Medically Attended Adverse Events (MAEs) and New Onset Chronic Diseases (NOCDs).
Description: A MAE was defined as any unsolicited symptom that received medical attention such as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. NOCDs included autoimmune diseases, diabetes mellitus.
Time Frame: From Day 0 to 182
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 78 | 152 | 151 | 151 | 148 | 50 | 50
Participants
  Subjects with MAEs | 16 | 29 | 33 | 28 | 34 | 14 | 14
  Subjects with NOCDs | 0 | 1 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 21-day follow-up period (Days 0-20) after vaccination.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 78 | 152 | 151 | 151 | 148 | 50 | 50
Participants | 30 | 67 | 60 | 73 | 84 | 26 | 20

8. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: as for outcome 7
Time Frame: Between Day 0 and Day 84 after vaccination.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 78 | 152 | 151 | 151 | 148 | 50 | 50
Participants | 35 | 77 | 71 | 81 | 89 | 29 | 23

9. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs).
Description: A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or resulted in a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to 182
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 78 | 152 | 151 | 151 | 148 | 50 | 50
Participants | 0 | 2 | 1 | 2 | 1 | 1 | 0

10. Secondary Outcome: Titers for Serum HI Antibodies Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 21 and Day 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 75 | 144 | 146 | 140 | 142 | 49 | 50
Titers
  H5N1 at Day 21 | 6.1 [5.2 to 7.1] | 22.5 [17.8 to 28.6] | 19.9 [15.7 to 25.3] | 23.5 [18.3 to 30.3] | 16.8 [13.5 to 20.9] | 23.0 [14.8 to 36.0] | 20.8 [13.9 to 31.3]
  H5N1 at Day 182: number analyzed (Participants) | 74 | 141 | 145 | 138 | 138 | 49 | 49
  H5N1 at Day 182 | 5.6 [5.1 to 6.2] | 27.8 [22.8 to 33.8] | 22.6 [18.4 to 27.9] | 26.1 [20.7 to 32.8] | 22.6 [18.3 to 28.0] | 32.5 [20.9 to 50.7] | 20.0 [13.6 to 29.3]

11. Secondary Outcome: Number of Seroconverted Subjects Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: as for outcome 1
Time Frame: At Days 21 and 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 75 | 144 | 146 | 140 | 142 | 49 | 50
Participants
  H5N1 at Day 21 | 5 | 60 | 60 | 64 | 54 | 23 | 21
  H5N1 at Day 182: number analyzed (Participants) | 74 | 141 | 145 | 138 | 138 | 49 | 49
  H5N1 at Day 182 | 2 | 77 | 66 | 67 | 62 | 24 | 23

12. Secondary Outcome: Geometric Mean Fold-rise (GMFR) Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: GMFR was defined as the geometric mean fold increase in serum HI antibody reciprocal titer on the specified study day compared to Day 0.
Time Frame: At Days 21 and 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 75 | 144 | 146 | 140 | 142 | 49 | 50
Fold increase
  H5N1at Day 21 | 1.2 [1.0 to 1.4] | 4.5 [3.6 to 5.7] | 4.0 [3.1 to 5.1] | 4.7 [3.6 to 6.0] | 3.3 [2.7 to 4.1] | 4.1 [2.7 to 6.2] | 4.2 [2.8 to 6.3]
  H5N1at Day 182: number analyzed (Participants) | 74 | 141 | 145 | 138 | 138 | 49 | 49
  H5N1at Day 182 | 1.1 [1.0 to 1.2] | 5.6 [4.6 to 6.8] | 4.5 [3.7 to 5.6] | 5.2 [4.1 to 6.5] | 4.5 [3.6 to 5.6] | 5.8 [3.7 to 9.1] | 4.0 [2.7 to 5.9]

13. Secondary Outcome: Number of Seroprotected Subjects Against the A/Indonesia/5/2005 (H5N1) Strain of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI antibody reciprocal titer ≥ 1:40 on the specified study day.
Time Frame: At Days 0, 21 and 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Number analyzed (Participants) | 75 | 144 | 146 | 140 | 143 | 49 | 50
Participants
  H5N1 at Day 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  H5N1 at Day 21: number analyzed (Participants) | 75 | 144 | 146 | 140 | 142 | 49 | 50
  H5N1 at Day 21 | 5 | 60 | 60 | 64 | 54 | 23 | 21
  H5N1 at Day 182: number analyzed (Participants) | 74 | 141 | 145 | 138 | 138 | 49 | 49
  H5N1 at Day 182 | 2 | 77 | 66 | 68 | 63 | 26 | 23

ADVERSE EVENTS:
Time Frame: Serious Adverse Events = From Days 0-182. Systematically assessed frequent adverse events (AEs) = During the 7 day post vaccination period. Non-systematically assessed frequent AEs= During Days 0-20 and Days 0-84 post vaccination period respectively.
Arm/Group | Pumarix Formulation 1 Group | Pumarix Formulation 2 Group | Pumarix Formulation 3 Group | Pandemrix Formulation A Group | Pandemrix Formulation B Group | Pumarix Formulation 4 Group | Pumarix Formulation 5 Group
Serious Adverse Events (participants affected / at risk) | 0/78 | 2/152 | 1/151 | 2/151 | 1/148 | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 45/78 | 137/152 | 132/151 | 146/151 | 131/148 | 48/50 | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pumarix Formulation 1 Group (N=78) | Pumarix Formulation 2 Group (N=152) | Pumarix Formulation 3 Group (N=151) | Pandemrix Formulation A Group (N=151) | Pandemrix Formulation B Group (N=148) | Pumarix Formulation 4 Group (N=50) | Pumarix Formulation 5 Group (N=50)
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pumarix Formulation 1 Group (N=78) | Pumarix Formulation 2 Group (N=152) | Pumarix Formulation 3 Group (N=151) | Pandemrix Formulation A Group (N=151) | Pandemrix Formulation B Group (N=148) | Pumarix Formulation 4 Group (N=50) | Pumarix Formulation 5 Group (N=50)
Pain (General disorders) | 18 | 133 | 130 | 139 | 124 | 48 | 42
Redness (General disorders) | 0 | 7 | 2 | 9 | 6 | 1 | 0
Swelling (General disorders) | 0 | 12 | 10 | 21 | 9 | 4 | 0
Fatigue (General disorders) | 16 | 64 | 50 | 67 | 69 | 15 | 15
Headache (General disorders) | 25 | 71 | 61 | 66 | 61 | 11 | 19
Joint pain (General disorders) | 12 | 49 | 36 | 53 | 39 | 11 | 11
Muscle aches (General disorders) | 15 | 74 | 64 | 86 | 63 | 19 | 21
Shivering (General disorders) | 4 | 18 | 21 | 27 | 17 | 8 | 6
Sweating (General disorders) | 6 | 23 | 12 | 24 | 21 | 5 | 1
Fever (General disorders) | 0 | 4 | 4 | 12 | 11 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 10 | 6 | 7 | 5 | 2 | 0 — Assessed within Days 0-20 following vaccination.
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 4 | 10 | 7 | 0 | 0 — Assessed within Days 0-20 following vaccination.
Headache (Nervous system disorders) | 3 | 3 | 3 | 13 | 12 | 4 | 4 — Assessed within Days 0-20 following vaccination.
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 2 | 5 | 7 | 2 | 4 — Assessed within Days 0-20 following vaccination.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 — Assessed within Days 0-20 following vaccination.
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 — Assessed within Days 0-20 following vaccination.
Nasopharyngitis (Infections and infestations) | 6 | 4 | 14 | 9 | 4 | 2 | 2 — Assessed within Days 0-84 following vaccination.
Headache (Nervous system disorders) | 3 | 4 | 3 | 13 | 12 | 4 | 4 — Assessed within Days 0-84 following vaccination.
Nausea (Gastrointestinal disorders) | 3 | 11 | 6 | 7 | 5 | 2 | 0 — Assessed within Days 0-84 following vaccination.
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 4 | 10 | 7 | 0 | 0 — Assessed within Days 0-84 following vaccination.
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 2 | 7 | 8 | 3 | 4 — Assessed within Days 0-84 following vaccination.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 — Assessed within Days 0-84 following vaccination.
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 — Assessed within Days 0-84 following vaccination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.